CLINICAL TRIAL: NCT06305650
Title: The Efficacy and Safety of a Probiotic in Reducing Body Fat and Blood Lipids Among Overweight and Obese Individuals
Brief Title: Probiotic Influence on Obesity-Related Lipidemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK2024001
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Overweight or Obesity
Keywords: Probiotic; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double（Participant,Investigator）
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): one bag/day BBr60, before meals
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Maltodextrin, one bag/day, before meals
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Through oral probiotic intervention for 12 weeks, participants' BMI, body fat percentage, and waist-to-hip ratio will be measured at weeks 0, 6, and 12, and fecal samples will be collected at weeks 0 and 12 for gut microbiota analysis.

SUMMARY:
This study aims to investigate the effects of Bifidobacterium breve BBr60 on key health indicators in overweight and obese adults. Specifically, it will assess the probiotic's impact on body composition metrics such as BMI, body fat percentage, WHR, and BMR. The inclusion criteria for participants are a BMI of ≥28 kg/m^2, targeting individuals who stand to benefit significantly from metabolic and body composition improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 28 kg/m2;
2. Voluntarily, in writing, and signing the informed consent form, agreeing to participate in this study;
3. Those who agree to abide by the protocol and study restrictions and are able to comply with a low-carbohydrate, energy-restricted diet plan.
4. Subjects (including male subjects) have no plans to have children from 14 days before screening to 6 months after the end of the trial and voluntarily take effective contraceptive measures;

Exclusion Criteria:

1. Taking items with similar functions to those tested in a short period of time will affect the judgment of the results;
2. Patients with severe allergies and immune deficiency;
3. Women who are pregnant, breastfeeding or planning to become pregnant;
4. Severe diseases of cardiovascular, lungs, liver, kidneys and other important organs, diabetes, thyroid disease, severe metabolic diseases, malignant tumors, and severe immune system diseases;
5. People who have used antibiotics in the past two weeks;
6. Those who failed to consume the test samples as required or failed to follow up on time, resulting in uncertainty in determining the efficacy;
7. Have used laxatives or fiber supplements in the past 6 weeks;
8. Subjects judged by other researchers to be unfit to participate. Those who meet any of the above conditions will not be selected.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Effect on body mass index (BMI) values. | 12 weeks
  After the probiotic intervention, the change in body mass index (BMI) from baseline in obese/overweight individuals will be calculated. BMI is measured by dividing a person's weight in kilograms by the square of their height in meters (kg/m^2).

CONTACTS AND LOCATIONS:
Locations (1):
- Henan University of Science and Technology, Luoyang, Henan, China